CLINICAL TRIAL: NCT01915914
Title: A Randomized, Open-label, Comparative Study to Evaluate an Intermittent Dosing Regimen of Fluticasone Propionate 0.05% Cream (Twice Per Week) in Reducing the Risk of Relapse When Added to Regular Daily Moisturization Using PHYSIOGEL Lotion in Paediatric Subjects With Stabilized Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117291
Record Dates: First submitted 2013-06-27; First posted 2013-08-05 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases | interventions — Fluticasone

ARMS (2):
- fluticasone propionate (Experimental): To evaluate an intermittent dosing regimen of fluticasone propionate 0.05% cream (twice per week) in reducing the risk of relapse when added to regular daily moisturization using PHYSIOGEL Lotion in paediatric subjects with stabilized atopic dermatitis
  Interventions: Drug: Fluticasone propionate
- physiogel (Active Comparator): To compare the efficacy and safety of fluticasone propionate 0.05% cream (twice per week) added to regular daily moisturization using Physiogel Lotion with Physiogel Lotion alone in paediatric subjects with stabilized atopic dermatitis
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Fluticasone propionate — All subjects receive FP 0.05% cream twice daily up to 4 weeks to all affected sites and any newly occurring sites in ACUTE phase. After randomization in MAINTENANCE phase, subjects either receive emollient (Physiogel) twice daily extendedly plus FP 0.05% cream once daily twice a week to all healed sites and any newly occurring sites (Group A), or emollient (Physiogel) twice daily extendedly (Group B), up to 20 weeks. In FOLLOW-UP phase, all subjects apply emollient (Physiogel) twice daily up to 12 weeks.

SUMMARY:
This is an open-label, randomized, comparative study, including 4 phases: SCREENING, ACUTE, MAINTENANCE and FOLLOW-UP.

Subjects will complete the SCREENING phase to check the eligibility within 7 days after they sign the written informed consent form. All eligible subjects will be enrolled in ACUTE phase to receive twice daily Fluticasone propionate (FP) 0.05% cream up to 4 weeks. The efficacy and safety in ACUTE phase will be assessed every 2 weeks up to 4 weeks or until Treatment Success which depends on which time point comes first. Then subject can get into the MAINTENANCE phase receiving either emollient twice daily plus FP 0.05% cream once daily twice a week (Group A), or emollient twice daily (Group B), by 1:1 randomization. The treatment duration in MAINTENANCE phase will be up to 20 weeks. The efficacy and safety in MAINTENANCE phase will be assessed every 4 weeks up to 20 weeks or until AD relapse that depends on which time point comes first. If subjects don't experience relapse during MAINTENANCE phase, subsequent FOLLOW-UP phase applying emollient twice daily won't be longer than another 12 weeks.

Total study duration is up to 37 weeks. All subjects receive FP 0.05% cream twice daily up to 4 weeks to all affected sites and any newly occurring sites in ACUTE phase. After randomization in MAINTENANCE phase, subjects either receive emollient twice daily extendedly plus FP 0.05% cream once daily twice a week to all healed sites and any newly occurring sites (Group A), or emollient twice daily extendedly (Group B), up to 20 weeks. In FOLLOW-UP phase, all subjects apply emollient twice daily up to 12 weeks.

This study will enrol 120 subjects, and propose at least 80 subjects to be randomized.

Study Endpoints/Assessments:

Primary endpoint is to observe the median time to the first relapse of AD during MAINTENANCE phase.

Secondary endpoints are:

1. Median time to the first relapse of AD during the whole study (including maintenance phase and follow-up phase.
2. Numbers of recurrent patients at the end of MAINTENANCE phase;
3. Numbers of recurrent patients at the end of FOLLOW-UP phase;
4. The effective rates (proportion of "treatment success" patients) during ACUTE phase (V3, W-2±2days;V4, W0±2days )
5. Evaluate the safety during the whole study duration (ACUTE phase, MAINTENANCE phase, FOLLOW-UP phase respectively);
6. Evaluate visual skin assessment for signs of cutaneous atrophy, epidermal thickening / lichenification and abnormal pigmentation changes during the whole study duration (ACUTE phase, MAINTENANCE phase, FOLLOW-UP phase respectively);
7. The change of Quality of Life (QoL) from baseline at the end of MAINTENANCE phase;
8. The change of Quality of Life (QoL) from baseline at the end of FOLLOW-UP phase;
9. Subjects' post-study evaluation to drugs.

DETAILED DESCRIPTION:
Background Atopic dermatitis (AD) is a chronic relapsing skin disease caused by the intervention of plural unspecific stimulation or specific allergens accompanied with cutaneous physiologic dysfunction. AD is one of the most common skin diseases which effects up to 20% of Children and 1-3% of adults in most of countries of the world. The data from a Chinese epidemiologic research shows the prevalence rate of AD is 10.9%in school-age adolescent and 15.3% in preschool children in 2010.

Around 65% patients with AD develop the symptoms in the first year of life; and 90% patients develop the symptoms before 5 years of age. Onset of atopic dermatitis in adolescence or later is uncommon.

The objective of treatment in AD is to relief symptoms and reduces the cutaneous inflammation. Emollients as the mainstay of maintenance therapy are able to restore skin barrier function. Topical glucocorticoids recommended as first line treatment are important anti-inflammatory drugs to be used in AD, especially in the acute phase.

One of the most troublesome features of AD is its chronic relapsing nature suggesting the need for a long-term therapy of this disease. The common long-term treatment of AD is a reactive treatment approach based on the daily application of emollients accompanied by the application of topical glucocorticoids (TCS) or calcineurin inhibitors (TCI) 'as needed'. However, a new alternative treatment 'proactive therapy' has been proven its effective and well-tolerated to reduce AD relapse in clinical trials and recommended by guidelines.

This proactive therapy starts with an intensive topical anti-inflammatory therapy until all lesions have virtually cleared, followed by long-term, low-dose intermittent application of anti-inflammatory drugs to previous affected and now clinically healthy-looking skin combined with daily application of emollients to always unaffected areas.

Latest Chinese guideline of AD recommends the application of emollients or moisturizers in both the acute and maintenance phase, and intermittent application of topical corticosteroids with daily use of emollients and moisturizers as the first-line option of AD therapy.

However, the concept of 'proactive therapy' of AD has not been well accepted by Chinese dermatologists. In context, the studies demonstrated 'proactive therapy' efficacy has been done mainly in Caucasian subjects instead of in Chinese population. For this reason, there still exist unmet medical needs to generate data on combination use of fluticasone propionate with moisturizer in AD maintenance therapy in China.

Rationale Fluticasone propionate (FP) is a synthetic fluorinated corticosteroid of medium strength for the topical treatment of skin disease. The established glucocorticoids showed anti-inflammatory, anti-proliferative and immunosuppressive effects. FP has been demonstrated havinga moderate anti-inflammatory effect associated with good compliance among patients, a low incidence of cross-sensitivity reactions and a weak atrophogenicity.

FP does not show a significant effect on the hypothalamic pituitary axis (HPA), due to its lipophilicity, and its rapid hepatic biotransformation, reflecting a favourable ratio between topical and systemic activity. The results from a clinical trial with moderate to severe AD demonstrate that FP does not cause any major local side-effect. First-line therapy of AD in paediatric patients consist of the application of a mildly to moderately potent topical glucocorticoid combined with emollients . FP cream 0.05% has also been proven safe for the treatment of moderate to severe AD for up to 4 weeks in children 3 months of age and older.

More than one study has been demonstrated the efficacy and safety of FP 0.05% cream for proactive therapy of AD. A large multicentre study compared an intermittent dosing regimen of FP 0.05% cream (twice per week) with its drug-free vehicle in reducing the risk of relapse in adults and children (44% and 66% respectively) aged 3 months to 65 years with moderate or severe, but stabilized AD. Both regimens were added to regular daily emollient. The results showed patients receiving intermittent FP cream in the maintenance phase were 7.7 times (paediatric patients even 8.1 times) less likely to have an AD relapse compared with patients under vehicle cream. And the maintenance therapy with FP turned out to be safe and well-tolerated.

Subsequent similar large scale study was to compare the efficacy and safety of both FP 0.05% cream and 0.005% ointment in reducing the risk of relapses. The difference was that only patients aged 12-65 years with moderate to severe AD who were experiencing a flare were enrolled. FP 0.05% was more effective in reducing relapses than FP 0.005%: the former reducing the risk of relapses six fold and the latter two fold compared with emollient alone. Median time to relapse was 6 weeks for emollient alone compared with more than 16 weeks for additional FP. Both medications were well-tolerated with a low risk of local adverse effects.

First-line therapy of AD in paediatric patients consist of the application of a mildly to moderately potent topical glucocorticoid combined with emollients . Except for topical glucocorticoid, emollients are the basic treatment of AD, which have been recommended and emphasized by almost all the AD guidelines. PHYSIOGEL lotion, as a hypoallergenic emollient, contains physiological lipids, which mimics the structure and composition of the skin's protective lipid barrier with DMS (Dermal Membrane Structure) technique. PHYSIOGEL lotion provides immediate and long lasting moisture to prevent skin dryness, which has been recommended by dermatologists in AD adjunctive daily care. It is advised to apply a thin film of PHYSIOGEL lotion once to twice daily ideally for people of all ages with dry, sensitive and barrier dysfunction skin (including people suffering from AD).

In summary, a superiority of a proactive therapy with combination of FP and emollient over the drug-free vehicle or emollient alone has been demonstrated. Proactive therapy with FP prevented, delayed, and reduced the occurrence of exacerbations and AD relapses without any obvious safety concerns. Besides, PHYSIOGEL lotion, an emollient with physiological lipids and DMS technology, has good efficacy in repairing skin barrier. In this regard, it is possibly meaningful to demonstrate the efficacy and safety of a FP and PHYSIOGEL lotion combination in reducing AD relapse.

OBJECTIVE(S) This study is aimed to demonstrate the risk of AD relapse can be significantly reduced by extended intermittent dosing with Fluticasone propionate (FP) 0.05% cream in addition to regular emollient therapy (PHYSIOGEL lotion) in the maintenance treatment (20 weeks) of atopic dermatitis (AD) as compared with application of emollient alone.

The secondary objective is to evaluate the safety of FP 0.05% cream and emollient combination usage in AD maintenance treatment and determine the optimal treatment regimen in Chinese paediatric patients with AD.

Study Design This is an open-label, randomized, comparative study. The study includes 4 phases: SCREENING, ACUTE, MAINTENANCE and FOLLOW-UP.

After subjects sign the written informed consent form (Visit 1), they will enter the SCREENING phase to check the eligibility within 7 days before the 1st dose of FP 0.05% cream. During SCREENING phase, investigator will collect subjects' demographic data, medical history, Atopic Dermatitis' diagnosis and treatment history, concomitant medications. Investigator needs to assess AD Severity and conduct physical examination. Substance abuse will be evaluated. And pregnant test must be conducted to check for Women of childbearing potential (WOCBP).

-Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study (and for up to 6 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal.

Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or here their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential.

The Visit 2 will be occurred before the 1st dose of FP 0.05% cream. At Visit 2, investigator needs to evaluate Eczema Area, AD Severity and Visual Skin Assessment. Vital signs will be measured and recorded. Subjects need to complete the questionnaire of QoL under the investigator's instruction. Investigator must confirm subjects' eligibility for ACUTE phase after all of inclusion and exclusion criteria have been checked.

All subjects eligible for ACUTE phase will receive twice daily FP 0.05% cream. FP 0.05% cream will be applied to affected sites and any newly occurring AD sites.

The efficacy and safety in ACUTE phase will be assessed every 2 weeks up to 4 weeks or until Treatment Success dependent on which time point comes first. At each visit (Visit 3, W-2±2days; Visit 4, W0±2days) in ACUTE phase, investigator needs to assess Eczema Area, AD Severity, Visual Skin Assessment, and conduct physical examination, vital sign measurement. Randomization will be processed once investigator confirms the subject's eligibility for MAINTENANCE phase.

The day of randomization is D0 in MAINTENANCE phase. If patients achieve Treatment Success and meet the criteria of MAINTENANCE phase during the visit intervals of ACUTE phase, Visit 4 can be moved earlier than scheduled date. If the time of treatment success is within 2 weeks after Visit 2, the subject can enter Visit 4 directly by skipping Visit 3.

If patients don't achieve Treatment Success for 4-week FP 0.05% cream treatment, they will be discontinued study treatment and conduct End of Therapy Visit. The subjects eligible for MAINTENANCE phase will be 1:1 randomized to receive either emollient twice daily plus FP 0.05% cream once daily twice a week (Group A), or emollient twice daily (Group B). FP 0.05% cream will be applied to all healed sites and any newly occurring sites.

The efficacy and safety in MAINTENANCE phase will be assessed every 4 weeks up to 20 weeks or until AD relapse dependent on which time point comes first. At each visit (V5, W4±2days; V6, W8±2days; V7, W12±2days; V8,W16±2days;V9,W20±2days), Investigator needs to evaluate Eczema Area, AD Severity, Visual Skin Assessment, and conduct physical examination, vital sign measurement. The questionnaire of QoL needs to be completed by subjects at the end of maintenance phase.

In MAINTENANCE phase, once subjects experience AD Relapse, they will be discontinued study treatment and conduct End of Therapy Visit.

On the contrary, if subjects don't experience relapse during MAINTENANCE phase, all of them will enter FOLLOW-UP phase applying emollient twice daily.

The efficacy and safety in FOLLOW-UP phase will be assessed every 4 weeks up to 12 weeks or until AD relapse dependent on which time point comes first. At each visit (V10, W24±5days; V11, W28±5days; V12, W32±5days), investigator needs to evaluate Eczema Area, AD Severity, Visual Skin Assessment, and conduct physical examination, vital sign measurement.In FOLLOW-UP phase, once subjects experience AD relapse, they will be discontinued study treatment and conduct End of Therapy Visit.

At End of Therapy Visit, investigator needs to evaluate Eczema Area, AD Severity, Visual Skin Assessment, and conduct physical examination, vital sign measurement. Subjects need to complete the questionnaire of QoL and Subjects' post-study evaluation to drug.

Subjects need to conduct Early Withdrawal Visit once they meet Withdrawal Criteria. At Early Withdrawal Visit, investigator needs to evaluate Eczema Area, AD Severity, Visual Skin Assessment, and conduct physical examination, vital sign measurement. Subjects need to complete the questionnaire of QoL and Subjects' post-study evaluation to drug.

At each study visit, concomitant medications will be collected after receiving subject's written informed consent form, and AEs should be collected and documented after the first dose of FP. For the female subjects who has experienced menarche, urine pregnant test need to be done when subjects enter the study and be repeated at the end of the entire study. If the result is positive, the subject will quit from the study. The treatment compliance will be evaluated at each visit after the 1st dose of FP 0.05% cream.

Total study duration is up to 37 weeks.

ELIGIBILITY:
Inclusion Criteria:

Specific information regarding warnings, precautions, contraindications, adverse events, and other pertinent information on the GSK investigational product or other study treatment that may impact subject eligibility is provided in the package insert of CUTIVATE and PHYSIOGEL Lotion.

Deviations from inclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential. Subjects eligible for enrolment in the study must meet all of the following criteria:

1. male or female patients age between 1 to 18 years old (including 1 year and excluding 18 years old);
2. Diagnose atopic dermatitis according to criteria of Williams;
3. Mild to moderate AD on the head/neck, trunk, upper limbs or lower limbs and PSGA scores 2-3;
4. The informed consent must be signed before any study specific tests or procedures are initiated;

   Subjects eligible for enrolment in the MAINTENANCE phase of the study must meet all of the following criteria:
5. Achieve treatment success after receiving Fluticasone propionate 0.05% cream twice daily up to 4 weeks in ACUTE phase

Exclusion Criteria:

Deviations from exclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.

Subjects meeting any of the following criteria must not be enrolled in the study:

Acute phase:

1. Dermatitis of only the face, feet or hands;
2. The involved area has exceeded 10% of the whole body area;
3. Diagnosed contact dermatitis at predilection sites of AD;
4. Atrophy, telangiectasia, extensive scarring lesions in the area or areas to be treated;
5. Had topical therapies including but not limit to calcineurin inhibitors (topical tacrolimus or topical pimecrolimus), corticosteroids, antihistamines within 14 days prior to screening;
6. Has accepted nonsteroidal immunosuppressants (eg cyclosporine, methotrexate), or ultraviolet light treatments including ultraviolet-A and ultraviolet-B, or systemic corticosteroids regardless administration by oral, intramuscular, or intravenous within 4 weeks prior to screening;
7. Pregnant or breast-feeding. Women of Childbearing Potential (WOCBP) with a positive urine pregnancy test performed within 7 days before the start of treatment;
8. Has immunocompromised disease (e.g. lymphoma, AIDS, Wiskott-Aldrich syndrome) or have a history of malignancy (including basal cell carcinoma, squamous cell carcinoma, melanoma);
9. Has open skin infections (bacterial, viral or fungal) if at the application site;
10. Has head lice or scabies;
11. Present with clinical conditions other than AD that may interfere with the valuation (e.g. generalized erythrodema, toxicoderma, acne, Netherton's Syndrome, psoriasis);
12. Require systemic therapy for the treatment of atopic dermatitis, or had systemic therapy including but not limit to antihistamines within 14 days prior to screening;
13. Has accepted any experimental or investigational drug or therapy within 6 weeks prior to screening;
14. Has known hypersensitivity to Fluticasone Propionate 0.05% cream, or PHYSIOGEL lotion, or relate drugs;
15. Non-compliance with general medical treatment, or are known to miss appointments, or don't intend to comply with the protocol for the duration of the study;
16. Drug abuse, mental dysfunction, or other factors limiting the subject's ability to cooperate fully with study-related procedures;
17. Know to be unreliable or may be unable to complete the study;
18. Any condition or prior/present treatment that would render the subject not eligible for the study;

    Maintenance phase:
19. Accepted topic therapies other than Fluticasone propionate 0.05% cream and emollients during the ACUTE phase;
20. Has active skin infection (bacterial, viral or fungal).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2013-12-23 (Actual); Primary Completion 2015-02-15 (Actual); Study Completion 2015-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- China (4):
  - GSK Investigational Site, Shenzhen, Guangdong
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number of enrolled participants n=123 in Acute Phase and n=107 in Maintenance Phase (ITT Population).
Pre-assignment Details: Eligible participants (par.) received twice daily (BID) fluticasone propionate 0.05% (FP) cream up to 4 weeks (wk) (in Acute Phase), then par. received (1:1) either emollient BID plus FP cream once daily (OD) twice a wk, or emollient BID up to 20 wk (Maintenance Phase). Par. who did not relapse received emollient BID up to 12 wk (Follow-up Phase).
Groups:
- FP 0.05% Cream: Participants who satisfied eligibility criteria received FP 0.05% cream BID up to 4 weeks. FP 0.05% cream was applied to affected sites and any newly occurring atopic dermatitis (AD) sites. Investigator assessed Eczema Area, AD Severity, Visual Skin Assessment, and conducted physical examination, vital sign measurement in the Acute Phase. The efficacy and safety in the Acute Phase was assessed every 2 weeks up to 4 weeks or until treatment success.
- Emollient Plus FP 0.05% Cream: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as participants with Physician Static Global Assessment (PSGA) <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). During the Maintenance Phase, the participants received emollient BID plus FP 0.05% cream OD twice a week up to 20 weeks. FP 0.05% cream was applied to all healed sites and any newly occurring sites. Emollient was applied before the application of FP 0.05% cream to the affected and unaffected areas.
- Emollient: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as PSGA <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID up to 20 weeks.
- Follow-up: Emollient: Participants who completed the study treatment in the Maintenance Phase in either treatment group without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks.
Period: Acute Phase
Arm/Group | FP 0.05% Cream | Emollient Plus FP 0.05% Cream | Emollient | Follow-up: Emollient
Started | 123 | 0 | 0 | 0
Completed-Not Entered Maintenance Phase | 4 | 0 | 0 | 0
Completed | 111 | 0 | 0 | 0
Not Completed | 12 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Accepted Other Topic Therapies | 1 | 0 | 0 | 0
Not completed — Not Achieved "treatment success" | 1 | 0 | 0 | 0
Not completed — Missing | 1 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | FP 0.05% Cream | Emollient Plus FP 0.05% Cream | Emollient | Follow-up: Emollient
Started | 0 | 54 | 53 | 0
Completed | 0 | 48 | 51 | 0
Not Completed | 0 | 6 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 4 | 1 | 0
Not completed — Missing | 0 | 1 | 0 | 0
Period: Follow-up Phase
Arm/Group | FP 0.05% Cream | Emollient Plus FP 0.05% Cream | Emollient | Follow-up: Emollient
Started | 0 | 0 | 0 | 66
Completed | 0 | 0 | 0 | 64
Not Completed | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: Participants who entered the Acute Phase received FP 0.05% cream BID up to 4 weeks. FP 0.05% cream was applied to the affected sites and any newly occurring atopic dermatitis (AD) sites. The efficacy and safety in the Acute Phase assessed every 2 weeks up to 4 weeks or until treatment success. Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as participants with physician static global assessment (PSGA) <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). During the Maintenance Phase, participants received emollient BID plus FP 0.05% cream OD twice a week, or emollient BID, up to 20 weeks. Participants who completed the study treatment in the Maintenance Phase in either treatment group without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks.
Arm/Group | Overall
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.8 (2.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 60
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 118
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Relapse of AD During the Maintenance Phase
Description: Time to the first relapse of AD is defined as the number of days from start of the FP treatment in Maintenance Phase until AD relapse. AD relapse is defined as participants with PSGA exacerbation score >=2 (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe) compared to PSGA score of treatment success during Acute Phase. Participants with treatment success are defined as participants with PSGA <=1; and the improvement >=2 compared to Baseline.
Time Frame: From the start of treatment up to Week 20 during the Maintenance Phase
Population: ITT Population: all participants who were randomized into the Maintenance Phase. Only participants available at the specified time point were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Days | NA [NA to NA] — Limited number of participants had AD relapse during the study; therefore, the Median and CI could not be provided. | 142.0 [50.0 to 150.0]
Statistical Analysis 1: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 13.4993, 95% CI 2-sided [4.1113 to 44.3250]

2. Secondary Outcome: Median Time to the First Relapse of AD During the Maintenance Phase and Follow-up Phase
Description: Median time to the first relapse of AD during the Maintenance Phase and Follow-up Phase is defined as the number of days from start of the FP treatment until AD relapse during the Maintenance Phase and Follow-up Phase. AD relapse is defined as participants with PSGA exacerbation score >=2 (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe) compared to PSGA score of treatment success during the Acute Phase.
Time Frame: From the start of treatment up to Week 32 during the Maintenance Phase and Follow-up Phase
Population: ITT Population. Only participants avilable at the specified time point were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Emollient Plus FP 0.05% Cream: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as participants with Physician Static Global Assessment (PSGA) <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID plus FP 0.05% cream OD twice a week up to 20 weeks. FP 0.05% cream was applied to all healed sites and any newly occurring sites. Emollient was applied before the application of FP 0.05% cream to the affected and unaffected areas.Participants who completed the study treatment in the Maintenance Phase without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks.
- Emollient: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as PSGA <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID, up to 20 weeks. Participants who completed the study treatment in the Maintenance Phase without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks.
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Days | NA [NA to NA] — Limited number of participants had AD relapse during the study; therefore, the Median and CI could not be provided. | 142.0 [50.0 to NA] — Limited number of participants had AD relapse during the study; therefore, the upper limit of CI could not be provided.
Statistical Analysis 1: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 4.9524, 95% CI 2-sided [2.4258 to 10.1105]

3. Secondary Outcome: Numbers of Recurrent Participants at the End of the Maintenance Phase (Week 20)
Description: The number of participants with AD recurrent/relapse at the end of Maintenance Phase is presented. AD relapse is defined as participants with PSGA exacerbation score >=2 (the six-point scale of PSGA: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe) compared to PSGA score of treatment success. Participants with treatment success is defined as participants with PSGA <=1; and the improvement >=2 compared to Baseline.
Time Frame: From Week 0 (or treatment success, if earlier) to Week 20
Population: ITT Population
Measure: Number; unit: Participants
Groups:
- Emollient Plus FP 0.05% Cream: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as participants with Physician Static Global Assessment (PSGA) <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID plus FP 0.05% cream OD twice a week up to 20 weeks. FP 0.05% cream was applied to all healed sites and any newly occurring sites. Emollient was applied before the application of FP 0.05% cream to the affected and unaffected areas.
- Emollient: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as PSGA <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID, up to 20 weeks.
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Participants | 3 | 30
Statistical Analysis 1: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Secondary Outcome: Numbers of Recurrent Participants at the End of the Follow-up Phase (Week 32)
Description: The number of participants with AD recurrent/relapse at the end of the Follow-up Phase is presented. AD relapse is defined as participants with PSGA exacerbation score >=2 (the six-point scale of PSGA: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe) compared to PSGA score of treatment success. Participants with treatment success is defined as participants with PSGA <=1; and the improvement >=2 compared to Baseline.
Time Frame: From Week 20 to Week 32
Population: ITT Population
Measure: Number; unit: Participants
Groups:
- Emollient Plus FP 0.05% Cream: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as participants with Physician Static Global Assessment (PSGA) <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID plus FP 0.05% cream OD twice a week up to 20 weeks. FP 0.05% cream was applied to all healed sites and any newly occurring sites. Emollient was applied before the application of FP 0.05% cream to the affected and unaffected areas. Participants who completed the study treatment in the Maintenance Phase without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks.
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Participants | 10 | 32
Statistical Analysis 1: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p < 0.0001, Chi-squared

5. Secondary Outcome: Number of Participants With "Treatment Success" During the Acute Phase
Description: The number of participants with "treatment success" during the Acute Phase is presented. Participants with treatment success are defined as participants with PSGA <=1; and the improvement >=2 (the six-point scale of PSGA: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe) compared to Baseline in the Acute Phase of the study.
Time Frame: From the start of treatment up to Visit 4 (Week 0) or treatment success (depends on which time point comes first)
Population: Enrolled Population: all participants who were enrolled into the Acute Phase of the study.
Measure: Number; unit: Participants
Arm/Group | FP 0.05% Cream
Number analyzed (Participants) | 123
Participants | 107

6. Secondary Outcome: Change From Baseline in Quality of Life (QoL) at the End of the Maintenance Phase
Description: Infant's Dermatitis Quality of Life Index (IDQOL) and Children's Dermatology Life Quality Index (CDLQI) were used to evaluate quality of life for participants of age between 1 to 16 years. IDQOL and CDLQI questionnaires were designed for infants (below the age of 4 years) and children (age 4 to age 16) with atopic dermatitis, respectively. The IDQOL and CDLQI were calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score in each questionnaire, the more quality of life is impaired. The change from Baseline in the QoL score is based on each questionnaire at the end of the Maintenance Phase and is calculated as the score at the end of the Maintenance Phase minus the Baseline score. Baseline is defined as QoL scores obtained at Visit 4 (end of Acute Phase). A QOL is equal to IDQOL if the age of a participant is < 4 years and it is equal to CDLQI if the age of a participant is between 4 and 16 years.
Time Frame: Baseline and Week 20
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Scores on a scale | -0.4 (4.40) | 2.2 (4.68)
Statistical Analysis 1: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p < 0.0001, ANCOVA

7. Secondary Outcome: Change From Baseline in QoL at the End of the Follow-up Phase
Description: Infant's IDQOL and Children's CDLQI were used to evaluate quality of life for participants of age between 1 to 16 years. IDQOL and CDLQI questionnaires were designed for infants (below the age of 4 years) and children (age 4 to age 16) with AD, respectively. The IDQOL and CDLQI were calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score in each questionnaire, the more quality of life is impaired. The change from Baseline in QoL score is based on each questionnaire at the end of the Follow-up Phase and is calculated as the score at the end of the Follow-up Phase minus the Baseline score. Baseline is defined as QoL scores obtained at Visit 4 (end of Acute Phase). A QOL is equal to IDQOL if the age of a participant is < 4 years and it is equal to CDLQI if the age of a participant is between 4 and 16 years.
Time Frame: Baseline and Week 32
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Emollient Plus FP 0.05% Cream: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as participants with Physician Static Global Assessment (PSGA) <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID plus FP 0.05% cream OD twice a week, up to 20 weeks. FP 0.05% cream was applied to all healed sites and any newly occurring sites. Emollient was applied before the application of FP 0.05% cream to the affected and unaffected areas.Participants who completed the study treatment in the Maintenance Phase without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks.
- Emollient: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as PSGA <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe).During the Maintenance Phase, the participants received emollient BID up to 20 weeks. Participants who completed the study treatment in the Maintenance Phase without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks.
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Scores on a scale | 0.0 (4.97) | 2.2 (5.10)
Statistical Analysis 1: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p < 0.0001, ANCOVA

8. Secondary Outcome: Number of Participants With Post-study Assessment of Skin Emollients Using Questionnaire
Description: Participants from each group completed the post-study questionnaire to rate the skin emollients (gel, lotion, cream, ointment, solution and foam) used in the past based on their experience. Participants rated skin emollients on a 5-point scale (5= "liked the best", 4= "second best", 3= "third best", 2= "fourth best, 1= "liked the least", N/A=Does not apply to me).
Time Frame: At early withdrawal or end of the therapy visit (up to Week 32)
Population: ITT Population
Measure: Number; unit: Participants
Groups:
- Emollient Plus FP 0.05% Cream: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as participants with Physician Static Global Assessment (PSGA) <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID plus FP 0.05% cream OD twice a weekup to 20 weeks. FP 0.05% cream was applied to all healed sites and any newly occurring sites. Emollient was applied before the application of FP 0.05% cream to the affected and unaffected areas. Participants who completed the study treatment in the Maintenance Phase without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks.
- Emollient: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as PSGA <=1; and the improvement >=2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). During the Maintenance Phase, the participants received emollient BID up to 20 weeks. Participants who completed the study treatment in the Maintenance Phase without a relapse, were entered into the Follow-up Phase. Emollient was applied BID up to 12 weeks to the affected and unaffected areas.
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Participants
  Gel, 1 | 2 | 1
  Gel, 2 | 2 | 1
  Gel, 3 | 2 | 2
  Gel, 4 | 2 | 2
  Gel, 5 | 1 | 0
  Gel, N/A | 39 | 44
  Lotion, 1 | 1 | 1
  Lotion, 2 | 0 | 1
  Lotion, 3 | 7 | 2
  Lotion, 4 | 8 | 12
  Lotion, 5 | 27 | 26
  Lotion, N/A | 5 | 8
  Cream, 1 | 1 | 0
  Cream, 2 | 1 | 2
  Cream, 3 | 7 | 2
  Cream, 4 | 12 | 18
  Cream, 5 | 6 | 5
  Cream, N/A | 21 | 23
  Ointment, 1 | 1 | 3
  Ointment, 2 | 7 | 3
  Ointment, 3 | 5 | 10
  Ointment, 4 | 3 | 3
  Ointment, 5 | 10 | 11
  Ointment, N/A | 22 | 20
  Solution, 1 | 0 | 1
  Solution, 2 | 1 | 0
  Solution, 3 | 4 | 5
  Solution, 4 | 4 | 2
  Solution, 5 | 1 | 0
  Solution, N/A | 38 | 42
  Foam, 1 | 4 | 2
  Foam, 2 | 1 | 1
  Foam, 3 | 1 | 0
  Foam, 4 | 0 | 0
  Foam, 5 | 0 | 0
  Foam, N/A | 42 | 47

9. Secondary Outcome: Number of Participants With Post-study Assessment of Lotion Qualities (1) Using Questionnaire
Description: Participants from each group completed the post-study questionnaire to rate the qualities of the lotion as compared with other skin emollients used in the past based on their experience. Each participant was asked the following Questions (Q). Q 1: This product is easier to use than other skin emollients; Q 2: When I apply this product I am able to start my daily activities quicker than with other skin emollients; Q 3: This product leaves my skin feeling softer than other skin emollients; Q 4: I am able to apply this product to larger body surface areas than other skin emollients; Q 5: This product disappears into my skin quicker than when I apply other skin emollients. Participants rated the qualities of the lotion based on a 5 point scale (5= "Strongly Agree", 4= "Agree", 3= "Neutral", 2= "Disagree", 1= "Strongly Disagree" N/A=Does not apply to me). Participant's rating for each question were summarized.
Time Frame: At early withdrawal or end of the therapy visit (up to Week 32)
Population: Enrolled Population
Measure: Number; unit: Participants
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Participants
  Q 1, 1 | 0 | 0
  Q 1, 2 | 0 | 4
  Q 1, 3 | 5 | 13
  Q 1, 4 or 5 | 39 | 29
  Q 1, N/A | 4 | 4
  Q 2, 1 | 0 | 1
  Q 2, 2 | 1 | 2
  Q 2, 3 | 5 | 13
  Q 2, 4 or 5 | 38 | 29
  Q 2, N/A | 4 | 5
  Q 3, 1 | 0 | 0
  Q 3, 2 | 1 | 3
  Q 3, 3 | 4 | 9
  Q 3, 4 or 5 | 39 | 34
  Q 3, N/A | 4 | 4
  Q 4, 1 | 0 | 1
  Q 4, 2 | 0 | 1
  Q 4, 3 | 6 | 7
  Q 4, 4 or 5 | 38 | 37
  Q 4, N/A | 4 | 4
  Q 5, 1 | 0 | 2
  Q 5, 2 | 0 | 2
  Q 5, 3 | 6 | 10
  Q 5, 4 or 5 | 38 | 32
  Q 5, N/A | 4 | 4

10. Secondary Outcome: Number of Participants With Post-study Assessment of Lotion Qualities (2) Using Questionnaire
Description: Participants from each group completed the post-study questionnaire to rate the qualities of the lotion as compared with other skin emollients used in the past based on their experience. Each participant was asked the following Questions (Q). Q 1: It leaves my skin feeling soft and smooth; Q 2: There is nothing left on my skin; Q 3: Does not feel greasy; Q 4: Disappears into my skin quickly after I put it on; Q 5: Easy to apply; Q 6: Fragrance-free; Q 7: Spreadability; Q 8: Lack of stickiness. Participants rated the qualities of the lotion based on a 5 point scale (5= "Strongly Agree", 4= "Agree", 3= "Neutral", 2= "Disagree", 1= "Strongly Disagree" N/A=Does not apply to me). Participant's rating for each question were summarized.
Time Frame: At early withdrawal or end of the therapy visit (up to Week 32)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Participants
  Q 1, 1 | 0 | 0
  Q 1, 2 | 1 | 1
  Q 1, 3 | 3 | 11
  Q 1, 4 or 5 | 44 | 37
  Q 1, N/A | 0 | 1
  Q 2, 1 | 0 | 0
  Q 2, 2 | 3 | 4
  Q 2, 3 | 1 | 8
  Q 2, 4 or 5 | 44 | 38
  Q 2, N/A | 0 | 0
  Q 3, 1 | 0 | 2
  Q 3, 2 | 3 | 3
  Q 3, 3 | 2 | 10
  Q 3, 4 or 5 | 43 | 35
  Q 3, N/A | 0 | 0
  Q 4, 1 | 0 | 2
  Q 4, 2 | 1 | 3
  Q 4, 3 | 2 | 7
  Q 4, 4 or 5 | 45 | 38
  Q 4, N/A | 0 | 0
  Q 5, 1 | 0 | 2
  Q 5, 2 | 1 | 1
  Q 5, 3 | 2 | 5
  Q 5, 4 or 5 | 45 | 42
  Q 5, N/A | 0 | 0
  Q 6, 1 | 0 | 0
  Q 6, 2 | 0 | 0
  Q 6, 3 | 1 | 5
  Q 6, 4 or 5 | 47 | 45
  Q 6, N/A | 0 | 0
  Q 7, 1 | 0 | 0
  Q 7, 2 | 1 | 0
  Q 7, 3 | 2 | 9
  Q 7, 4 or 5 | 45 | 41
  Q 7, N/A | 0 | 0
  Q 8, 1 | 0 | 2
  Q 8, 2 | 3 | 3
  Q 8, 3 | 2 | 10
  Q 8, 4 or 5 | 43 | 35
  Q 8, N/A | 0 | 0

11. Secondary Outcome: Change From Baseline in Cutaneous Atrophy Sign Score, Epidermal Thickening /Lichenification Sign Score and Abnormal Pigmentation Score Using Visual Analogue Scale (VAS) at the End of the Acute Phase
Description: Investigator evaluated and scored the signs of cutaneous atrophy (CA), epidermal thickening/lichenification (ET/L) and abnormal pigmentation (AP) using Visual Analogue Scale (ranging from 0 to 10, higher values represent a worse outcome) based on their subjective judgment. The change from Baseline in each signs (Cutaneous atrophy, epidermal thickening / lichenification and abnormal pigmentation) score at the end of the Acute Phase (Visit 4 [Week 0 or treatment success, depend on which time point comes first) ±2day]) and is calculated as the score at Visit 4 minus the Baseline score. Baseline is defined as the VAS score for each sign obtained before the first dose of study drug in the Acute Phase of the study (Visit 2). Summation of the VAS scores for each sign (CA, ET/L and AP) was done to calculate the Total VAS score (ranging from 0 to 30, higher values represent a worse outcome) at Visit 4 of the Acute Phase of the study.
Time Frame: From the start of treatment up to Visit 4 (Week 0) or treatment success (depends on which time point comes first)
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | FP 0.05% Cream
Number analyzed (Participants) | 123
Scores on a scale
  Visit 4, CA | -0.3 (1.12)
  Visit 4, ET/L | -1.9 (1.57)
  Visit 4, AP | -0.7 (1.47)
  Visit 4, Total VAS Score | -2.9 (3.14)

12. Secondary Outcome: Change From Baseline in Cutaneous Atrophy Sign Score, Epidermal Thickening /Lichenification Sign Score and Abnormal Pigmentation Score Using Visual Analogue Scale (VAS) at the End of the Maintenance Phase and Follow-up Phase
Description: Investigator evaluated and scored the signs of cutaneous atrophy (CA), epidermal thickening/lichenification (ET/L) and abnormal pigmentation (AP) using the Visual Analogue Scale (ranging from 0 to 10, higher values represent a worse outcome) based on their subjective judgment. The change from Baseline in each sign (Cutaneous atrophy, epidermal thickening / lichenification and abnormal pigmentation) score at the end of the Maintenance Phase and Follow-up Phase and is calculated as the score at the end of the Maintenance and Follow-up Phase minus the Baseline score. Baseline is defined as VAS score for each sign obtained at Visit 4 (end of Acute Phase). Summation of VAS scores for each sign (CA, ET/L and AP) was done to calculate the Total VAS score (ranging from 0 to 30, higher values represent a worse outcome) at the Maintenance and Follow-up phase of study. The missing value was imputed using last-observation-carry-forward (LOCF) method.
Time Frame: Baseline, Week 20 and Week 32
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Emollient Plus FP 0.05% Cream | Emollient
Number analyzed (Participants) | 54 | 53
Scores on a scale
  Week 20, CA | -0.1 (0.44) | -0.2 (1.01)
  Week 20, ET/L | -0.4 (1.49) | 0.5 (1.51)
  Week 20, AP | -0.4 (1.42) | 0.0 (1.32)
  Week 32, CA | -0.1 (0.58) | -0.2 (1.03)
  Week 32, ET/L | 0.1 (1.19) | 0.6 (1.53)
  Week 32, AP | -0.3 (1.23) | 0.0 (1.35)
  Week 20, Total VAS Score | -0.9 (2.61) | 0.3 (2.75)
  Week 32, Total VAS Score | -0.3 (2.09) | 0.4 (2.82)
Statistical Analysis 1: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p = 0.7010, Wilcoxon (Mann-Whitney) — Week 20, CA
Statistical Analysis 2: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p = 0.0042, Wilcoxon (Mann-Whitney) — Week 20, ET/L
Statistical Analysis 3: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p = 0.0810, Wilcoxon (Mann-Whitney) — Week 20, AP
Statistical Analysis 4: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p = 0.2799, Wilcoxon (Mann-Whitney) — Week 32, CA
Statistical Analysis 5: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p = 0.1375, Wilcoxon (Mann-Whitney) — Week 32, ET/L
Statistical Analysis 6: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p = 0.1100, Wilcoxon (Mann-Whitney) — Week 32, AP
Statistical Analysis 7: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p = 0.0394, Wilcoxon (Mann-Whitney) — Week 20, Total VAS Score
Statistical Analysis 8: Comparison: Emollient Plus FP 0.05% Cream vs Emollient; Test type: Superiority or Other; p = 0.2237, Wilcoxon (Mann-Whitney) — Week 32, Total VAS Score

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study drug until follow-up (last dose of study treatment (emollient), up to Week 32).
Description: SAEs and non-serious AEs were collected in participants of the Safety Population, comprised of all participants who received study therapy during the Acute Phase, Maintenance Phase and Follow-up Phase and have a safety assessment in the Acute Phase, Maintenance Phase and Follow-up Phase of the study.
Groups:
- FP 0.05% Cream: Participants who satisfied eligibility criteria received FP 0.05% cream BID up to 4 weeks. FP 0.05% cream was applied to affected sites and any newly occurring atopic dermatitis (AD) sites. Investigator assessed Eczema Area, AD Severity, Visual Skin Assessment, and conducted physical examination, vital sign measurement in the Acute Phase. The efficacy and safety of FP 0.05% cream was assessed every 2 weeks up to 4 weeks or until treatment success.
- Emollient Plus FP 0.05% Cream: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as participants with Physician Static Global Assessment (PSGA) less than or equal to 1; and the improvement greater than or equal to 2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). During the Maintenance Phase, the participants received emollient BID plus FP 0.05% cream OD twice a week up to 20 weeks. FP 0.05% cream was applied to all healed sites and any newly occurring sites. Emollient was applied before the application of FP 0.05% cream to the affected and unaffected areas.
- Emollient: Participants with treatment success during the Acute Phase were enrolled in the Maintenance Phase. Treatment success is defined as PSGA less than or equal to 1; and the improvement greater than or equal to 2 compared to Baseline (the six-point scale of PSGA score range from 0 to 5 where 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe). The participants received emollient BID up to 20 weeks.
Arm/Group | FP 0.05% Cream | Emollient Plus FP 0.05% Cream | Emollient | Follow-up: Emollient
Serious Adverse Events (participants affected / at risk) | 0/116 | 2/53 | 0/53 | 0/66
Other Adverse Events (participants affected / at risk) | 4/116 | 9/53 | 9/53 | 11/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FP 0.05% Cream (N=116) | Emollient Plus FP 0.05% Cream (N=53) | Emollient (N=53) | Follow-up: Emollient (N=66)
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0 | 0
Mycoplasma infection (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FP 0.05% Cream (N=116) | Emollient Plus FP 0.05% Cream (N=53) | Emollient (N=53) | Follow-up: Emollient (N=66)
Nasopharyngitis (Infections and infestations) | 2 | 3 | 3 | 3
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2
Exanthema subitum (Infections and infestations) | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 4 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.